CLINICAL TRIAL: NCT00923884
Title: Prospective Analysis of Genotypes in Adults Undergoing Therapy for Lung Cancer
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090103; 09-C-0103
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2018-04-20

CONDITIONS: Carcinoma, Non-Small Cell Lung; Carcinoma, Small-Cell Lung
Keywords: NSCLC; Genotype; SCLC; Lung Cancer; Non-Small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

* The Lung Cancer section of the National Cancer Institute s Medical Oncology Branch is running a study to better understand which genes might be important in patients who are undergoing therapy for lung cancer.

Objectives:

* To find out if differences (also called polymorphisms) in specific genes lead to differences in outcomes (such as treatment success and survival rates) for patients who have been diagnosed with lung cancer.
* To establish a repository of genetic information for future studies of these differences and their relation to lung cancer.

Eligibility:

* Any individual who has been diagnosed with lung cancer and is being treated through the National Cancer Institute.

Design:

* After entrance in this study, patients will provide information to the researchers on age, gender, race/ethnicity, treatments received and response to treatments, and other specific information about their disease. This information will be kept confidential.
* Approximately half a tablespoon of blood will be drawn.
* Patients will be treated for lung cancer with normal treatment methods, as if they had not been enrolled in the study
* Some patients may be offered the option of enrolling in separate research protocols for cancer treatment, involving chemotherapy, surgery, or radiation.

DETAILED DESCRIPTION:
Background:

* Lung cancer is the leading cause of cancer deaths among men and women worldwide.
* Despite modern surgical, radiation, and chemotherapeutic interventions, the prognosis for patients with lung cancer remains poor, with an overall cure rate of less than 15%.
* Genetic polymorphisms in drug-metabolizing enzymes, transporters, growth factor and hormonal receptors, DNA repair enzymes, and transcription factors might affect an individual s response to chemotherapy and radiation.
* Interindividual differences in efficacy and toxicity of cancer chemotherapy and radiation are especially important given the narrow therapeutic index of these modalities.
* Many of these differences have not been extensively explored in patients with lung cancer.

Objectives:

* To better understand the genotype-phenotype relationship between genetic polymorphisms and clinical outcomes, with a focus on overall survival, following lung cancer therapy.
* To better understand differences in outcome between Caucasian and African American patients being treated for lung cancer as a function of genotype.
* To establish a DNA repository for the investigation of polymorphisms related to outcomes in lung cancer.
* To develop methodology for the isolation, enumeration and live cell culture of circulating tumor cells (CTC) from lung cancer patients with microfiltration devices.

Eligibility:

- All individuals with the diagnosis of lung cancer being treated at the Washington D.C. Veterans Affairs Medical Center or the Medical Oncology Branch of the National Cancer Institute (NCI).

Design:

* A single 7-ml sample of venous blood will be obtained from all patients enrolled onto this study, for isolation of DNA.
* Two 5 ml samples of venous blood, drawn immediately following the 7 ml sample, will be obtained from all patients enrolled on this study at the NCI Clinical Center (only), for CTC studies.
* Polymorphisms in the following genes: ABCB1, ABCG2, COMT, CYP17, CYP19, CYP1B1, CYP1A1, CYP1A2, CYP2C8, CYP2C9, CYP2J2, CYP3A4, CYP3A5, DPYD, EPHX2, ERalpha, ERbeta, ERCC1, ERCC2, GSTP1, HIF1A, MPO, MTHFR, NQO1, p53, PPARD, SLCO1B3, TYMS, UGT1A1, VEGF, VEGFR, EGFR, SLC28A1, CDA, XRCC1, OCT1, OCT2, CHRNA3 and CHRNA5 will be analyzed by the Clinical Pharmacology Program.
* Methodology for the isolation, enumeration, and live cell culture of CTC with microfiltration devices will be developed by the NCI Genetics Branch.
* Patients will be followed at the medical oncology clinic at the Washington DC VA Medical Center or the NCI and the following information will be recorded in a confidential database: age, gender, race/ethnicity, smoking history, histology, stage, treatment(s) received, response, toxicity, time to disease progression, time to death.
* Associations between genetic polymorphisms and response to therapy, toxicity and clinical outcomes will be analyzed.
* The results of the CTC studies will be applied to the initial development and clinical

validation of CTC technology and lung cancer assays.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients 18 years of age and older are eligible.
  2. Histologic diagnosis of primary lung carcinoma. For non small cell lung cancer, patients can be stage I to IV, and receive any treatment (surgical resection, chemotherapy, radiation, molecularly targeted therapy). For small cell lung cancer, patients can be limited or extensive stage and receive any treatment (surgical resection, chemotherapy, radiation, molecularly targeted therapy).
  3. Patients must have a performance status of ECOG 0, 1, 2, or 3 for admission to this protocol.
  4. Patients with a current diagnosis of or a prior history of other cancers may be included onto this protocol.
  5. Patients may have either normal organ function or impaired organ function.

EXCLUSION CRITERIA:

1. Children will not be eligible.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2009-03-18; Study Completion 2018-04-20

PRIMARY OUTCOMES:
Evaluation of the association between polymorphisms in the enzymes ABCB1, CYP1B1, and CYP19 and clinical outcomes, with overall survival of greatest interest, in patients undergoing treatment for lung cancer. | Death or the conclusion of a 5-year follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Arriagada R, Bergman B, Dunant A, Le Chevalier T, Pignon JP, Vansteenkiste J; International Adjuvant Lung Cancer Trial Collaborative Group. Cisplatin-based adjuvant chemotherapy in patients with completely resected non-small-cell lung cancer. N Engl J Med. 2004 Jan 22;350(4):351-60. doi: 10.1056/NEJMoa031644. PMID 14736927
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875